CLINICAL TRIAL: NCT01545960
Title: Scanning Kelvin Probe Measurements of Acupuncture Point
Brief Title: Evaluating Acupuncture Points With Scanning Kelvin Probe
Status: Suspended | Type: Observational
Why Stopped: Adjusting minor software glitches
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Andrew A. Ahn, Assistant Professor, Massachusetts General Hospital
Other Study IDs: 5R21AT005249-03 (NIH)
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Healthy Individuals; Acupuncture Points; Electrical Potential

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Volunteers
  Interventions: Other: not applicable in this study

INTERVENTIONS:
Other: not applicable in this study — No actual interventions will be administered for this study.

SUMMARY:
The purpose of this study is to characterize the surface electrical potential of acupuncture points with a Scanning Kelvin Probe.

DETAILED DESCRIPTION:
Acupuncture points are anatomical structures described by traditional Chinese medicine. To this day, however, their scientific and Western anatomical characterizations remain unclear. Past studies have suggested that acupuncture points are distinct electrically (increased electrical conductivity). To evaluate this claim, this study uses a Scanning Kelvin Probe to study the electrical potential of three acupuncture points and their respective adjacent controls in 24 healthy individuals. The Scanning Kelvin Probe is a novel device that measures the electrical potential of skin without actually touching the skin surface.

ELIGIBILITY:
Inclusion Criteria:

* Individuals without chronic medical condition requiring daily medications (hypertension, diabetes, hypothyroidism, etc).

Exclusion Criteria:

* Individuals with autonomic disorders (sweating irregularities), skin disorders, extensive burns/scars on the hand, tremors, neuromuscular conditions, restless leg syndrome, movement disorders, and implanted cardiac defibrillator/pacemaker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Electrical Potential at Acupuncture points | One day
  Scanning Kelvin Probe measurements of electrical potentials at 3 predetermined acupuncture points.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew C. Ahn, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital - Martinos Center for Biomedical Imaging, Charlestown, Massachusetts, United States